CLINICAL TRIAL: NCT03620643
Title: Phase II Study of ROS1 Targeting With Crizotinib in Advanced E-cadherin Negative, ER Positive Lobular Breast Cancer, Diffuse Gastric Cancer, Triple Negative Lobular Breast Cancer or CDH1-mutated Solid Tumours
Brief Title: Crizotinib in Lobular Breast, Diffuse Gastric and Triple Negative Lobular Breast Cancer or CDH1-mutated Solid Tumours
Acronym: ROLo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pfizer (Industry); Breast Cancer Now (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CCR4684
Record Dates: First submitted 2018-05-04; First posted 2018-08-08 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Lobular Breast Carcinoma; Gastric Cancer; Triple Negative Breast Cancer; CDH1 Gene Mutation
Keywords: Advanced E-cadherin negative gastric cancer; Oestrogen receptor positive lobular breast cancer; Crizotinib; Fulvestrant
MeSH Terms: conditions — Carcinoma, Lobular; Stomach Neoplasms; Triple Negative Breast Neoplasms | interventions — Crizotinib; Fulvestrant; Drugs, Generic

STUDY DESIGN:
Intervention Model Description: This multi-centre study design will aim to complete recruitment over 18 months from six high volume centres including the Royal Marsden. Parallel recruitment to breast and basket cancer cohorts will take place for this study.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Crizotinib Oral Capsule [Xalkori] monotherapy (Active Comparator): Arm 1 - Basket cohort (n=29 participants) were treated with Crizotinib Oral Capsule [Xalkori] (250 mg b.d) taken as monotherapy on a continuous dosing schedule. One treatment cycle for Crizotinib is 28 days long.
  Interventions: Drug: Crizotinib Oral Capsule [Xalkori]
- Crizotinib Oral Capsule [Xalkori] plus Fulvestrant injection (Active Comparator): Arm 2 - Lobular Breast Cancer cohort (n=29 participants) were treated with combination therapy. The combination therapy included; Crizotinib Oral Capsule [Xalkori] (250mg b.d.) plus Fulvestrant 50 mg/mL Prefilled Syringe [Faslodex or generic] intramuscular (IM) injection (500 mg per 1 cycle (q28 days, plus loading dose on day 15).
  Interventions: Drug: Crizotinib Oral Capsule [Xalkori]; Drug: Fulvestrant 50 MG/ML Prefilled Syringe [Faslodex or generic]

INTERVENTIONS:
Drug: Crizotinib Oral Capsule [Xalkori] — Crizotinib 250 mg Crizotinib 200mg
  Other Names: Xalkori
Drug: Fulvestrant 50 MG/ML Prefilled Syringe [Faslodex or generic] — Fulvestrant (Faslodex or generic) is supplied as two 5-mL clear neutral glass (Type 1) barrels, each containing 250mg/5mL of fulvestrant solution for intramuscular injection and fitted with a tamper evident closure.
  Other Names: Faslodex
  Arms: Crizotinib Oral Capsule [Xalkori] plus Fulvestrant injection

SUMMARY:
The purpose of this study was to find out how effective the combination of crizotinib and fulvestrant was in shrinking lobular breast cancer tumours. The investigators also assessed the side effects of the combination of crizotinib tablets and fulvestrant injections. The side effects and the doses of crizotinib and fulvestrant had already been evaluated in large clinical trials, but this was the first time these two drugs had been combined together.

DETAILED DESCRIPTION:
This clinical study was looking at whether a drug called crizotinib, which is used in some patients with lung cancer, was effective in a sub-type of breast cancer, called lobular breast cancer. As the majority of lobular breast cancers are oestrogen receptor positive (ER+ve), crizotinib was combined with a second drug, fulvestrant, to try to block tumour growth that is driven by oestrogen.

Crizotinib targets cancers with genetic changes in two genes called ALK and ROS1. Lung cancers with changes in these genes usually get smaller when treated with crizotinib. Laboratory work at the Institute of Cancer Research has shown that lobular breast cancer cells, due to a mutation in a different gene called CDH1, appear to be similarly affected by crizotinib.

Fulvestrant is an oestrogen receptor down regulator and blocks the effects of oestrogen on oestrogen receptor positive (ER+ve) breast cancer cells. Fulvestrant is an established and approved anti-hormone therapy which patients with breast cancers are receiving in the clinic. It is possible that the combination of crizotinib and an anti-oestrogen agent will shrink the tumour(s) more effectively and prevent further growth. Because fulvestrant is only effective in post-menopausal women, if participants had not yet gone through the menopause, participants needed to start (or continue to receive) a monthly injection under the skin to temporarily stop the function of the participant's ovaries to be eligible to take part in the trial.

This injection is called goserelin and had to be started at least 4 weeks before the first day of treatment on the trial.

The overall aims of this clinical study were to find out:

* The proportion of patients whose tumour(s) shrink when they are treated with crizotinib and fulvestrant
* The safety and tolerability of fulvestrant in combination with crizotinib, to determine that they can be given together without unacceptable side effects
* What the drugs do to the tumours, which will help us decide which patients may benefit from this combination in the future

ELIGIBILITY:
Inclusion Criteria:

- Patients with histological diagnosis of E-cadherin negative inoperable or metastatic diffuse gastric cancer (basket cohort), Or inoperable or metastatic triple negative lobular breast cancer (basket cohort) Or inoperable or metastatic CDH1-mutated solid tumour with allele fraction ≥20% (basket cohort) Or recurrent inoperable locally advanced ER positive/HER2 negative lobular breast cancer (breast cohort).

Assessment of E-cadherin, ER and HER2 status as per local assessment.

- Lobular breast cancer patients previously treated with at least one prior line of therapy including at least one prior line of hormone therapy for advanced disease, but no more than three prior lines of chemotherapy for advanced disease.

Gastric cancer, triple negative lobular breast cancer or CDH1-mutated solid tumour patients previously treated with at least one prior therapy for advanced disease OR relapsing within one year of completing (neo) adjuvant chemotherapy OR unsuitable for chemotherapy in the opinion of the investigator (for example patient choice not to have chemotherapy, or no suitable chemotherapy agent).

* Measurable disease (RECIST 1.1)
* Haematological and biochemical indices within the ranges shown in protocol. These measurements must be performed within one week (Day -7 to Day 1) before the patient goes in the trial.
* Female patients with child-bearing potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial. Both male and female patients of reproductive potential must agree to use two forms of highly effective contraception (see below) for 2 weeks before starting the study treatment, throughout the treatment period and for 90 days after discontinuation of treatment with crizotinib and 2 years after the last dose of fulvestrant.

NOTE: it is only considered highly effective if the patient is refraining from sexual intercourse during the entire period of risk associated with the study treatments

The oral contraceptive pill may be ineffective when taken with crizotinib so is not an acceptable means of contraception for female patients during this study but can be used by female partners of male patients.

* 18 years of age or over with written (signed and dated) informed consent and be capable of co-operating with treatment and follow-up.
* World Health Organisation (WHO) performance status 0,1 or 2
* Estimated life expectancy of at least 3 months in the opinion of the investigator
* Pre-/peri-menopausal ER+ lobular breast cancer patients must be willing to receive gosarelin injections every 28 days.
* Signed and dated informed consent.
* Patients willing and able to comply with scheduled visits, treatment plans, laboratory tests, and other procedures.

Exclusion Criteria:

* Systemic chemotherapy or investigational medicinal products during the previous four weeks, or hormonal therapy within 7 days except luteinizing hormone-releasing hormone (LHRH) analogues for ovarian suppression. Bisphosphonates or RANK ligand antagonists are permitted for the management of bone metastases.
* Previous treatment with any agent that inhibits ROS1
* Mixed ductal/lobular breast cancer, unless both ductal and lobular components are CDH1 negative by local assessment
* Major surgery (excluding minor procedures, e.g. placement of vascular access) within 4 weeks or radiation therapy within 14 days prior to study entry
* Patients with known symptomatic brain metastases requiring steroids, untreated brain metastases or spinal cord compression
* Any of the following within 12 months prior to study entry: myocardial infarction, uncontrolled angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack. Uncontrolled hypertension or cardiac dysrhythmia including atrial fibrillation.
* QT interval, corrected >470 ms or the use of bradycardic agents, drugs which prolong the QT interval and/or anti-arrhythmic agents within 12 days before the first dose of crizotinib or during study treatment.
* Use of drugs that are known potent cytochrome P450 (CYP) 3A4 inhibitors or moderate or strong CYP 3A4 inducers within 12 days before the first dose of crizotinib. Us of CYP3A4 substrates with a narrow therapeutic index (such as ciclosporin) is also not permitted within 12 days prior or during the study treatment.
* Patients on warfarin. Patients requiring anticoagulation for rate-controlled AF or previous venous thromboembolism should be switched to low-molecular weight heparin.
* Known HIV or AIDS-related illness, active infection requiring systemic therapy, or positive HBV or HCV test indicating acute or chronic infection.
* Inability or unwillingness to swallow pills, or (for patients receiving fulvestrant) receive IM injections.
* Other severe acute or chronic medical condition or psychiatric condition, recent or active suicidal ideation or behaviour, or end stage renal disease on haemodialysis, or laboratory abnormality that may increase the risk associated with study participation or investigational products administration or may interfere with the interpretation of results and, in the judgment of the Investigator, would make the patient inappropriate study entry.
* Persisting toxicity related to prior therapy >Grade 1 (except for stable peripheral neuropathy grade ≤2 or alopecia grade ≤2).
* Pregnancy or lactation.
* Diagnosis of other malignancy within 5 years, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the breast or cervix, or low-grade (Gleason ≤6) prostate cancer.
* Is a participant or plans to participate in another interventional clinical trial, whilst taking part in this study. Participation in an observational trial would be acceptable.
* Immunocompromised status due to current known active infection with HIV or due to the use of immunosuppressive therapies for other conditions
* Known prior or suspected hypersensitivity to investigational products or to any of the excipients.
* Patients at risk for gastrointestinal perforation (due to e.g., history of diverticulitis).
* Any other condition which in the Investigator's opinion would not make the patient a good candidate for the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-09 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Peter Schmid, Study Chair — St Bart's Hospital
Locations (5):
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Royal Marsden NHS Foundation Trust, London
  - Guys and St Thomas NHS Foundation Trust, London
  - University College London Hospital, London
  - The Christie NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Christgen M, Derksen P. Lobular breast cancer: molecular basis, mouse and cellular models. Breast Cancer Res. 2015 Feb 8;17(1):16. doi: 10.1186/s13058-015-0517-z. PMID 25757734
- [Background] Jeanes A, Gottardi CJ, Yap AS. Cadherins and cancer: how does cadherin dysfunction promote tumor progression? Oncogene. 2008 Nov 24;27(55):6920-9. doi: 10.1038/onc.2008.343. PMID 19029934
- [Background] Bertucci F, Orsetti B, Negre V, Finetti P, Rouge C, Ahomadegbe JC, Bibeau F, Mathieu MC, Treilleux I, Jacquemier J, Ursule L, Martinec A, Wang Q, Benard J, Puisieux A, Birnbaum D, Theillet C. Lobular and ductal carcinomas of the breast have distinct genomic and expression profiles. Oncogene. 2008 Sep 11;27(40):5359-72. doi: 10.1038/onc.2008.158. Epub 2008 May 19. PMID 18490921
- [Background] Cristofanilli M, Gonzalez-Angulo A, Sneige N, Kau SW, Broglio K, Theriault RL, Valero V, Buzdar AU, Kuerer H, Buchholz TA, Hortobagyi GN. Invasive lobular carcinoma classic type: response to primary chemotherapy and survival outcomes. J Clin Oncol. 2005 Jan 1;23(1):41-8. doi: 10.1200/JCO.2005.03.111. PMID 15625359
- [Background] Graziano F, Humar B, Guilford P. The role of the E-cadherin gene (CDH1) in diffuse gastric cancer susceptibility: from the laboratory to clinical practice. Ann Oncol. 2003 Dec;14(12):1705-13. doi: 10.1093/annonc/mdg486. PMID 14630673
- [Background] Pernot S, Voron T, Perkins G, Lagorce-Pages C, Berger A, Taieb J. Signet-ring cell carcinoma of the stomach: Impact on prognosis and specific therapeutic challenge. World J Gastroenterol. 2015 Oct 28;21(40):11428-38. doi: 10.3748/wjg.v21.i40.11428. PMID 26523107
- [Background] Peng Z, Li Z, Gao J, Lu M, Gong J, Tang ET, Oliner KS, Hei YJ, Zhou H, Shen L. Tumor MET Expression and Gene Amplification in Chinese Patients with Locally Advanced or Metastatic Gastric or Gastroesophageal Junction Cancer. Mol Cancer Ther. 2015 Nov;14(11):2634-41. doi: 10.1158/1535-7163.MCT-15-0108. Epub 2015 Sep 1. PMID 26330547
- [Background] Turner N, Grose R. Fibroblast growth factor signalling: from development to cancer. Nat Rev Cancer. 2010 Feb;10(2):116-29. doi: 10.1038/nrc2780. PMID 20094046
- [Background] Solomon BJ, Mok T, Kim DW, Wu YL, Nakagawa K, Mekhail T, Felip E, Cappuzzo F, Paolini J, Usari T, Iyer S, Reisman A, Wilner KD, Tursi J, Blackhall F; PROFILE 1014 Investigators. First-line crizotinib versus chemotherapy in ALK-positive lung cancer. N Engl J Med. 2014 Dec 4;371(23):2167-77. doi: 10.1056/NEJMoa1408440. PMID 25470694
- [Background] Shaw AT, Ou SH, Bang YJ, Camidge DR, Solomon BJ, Salgia R, Riely GJ, Varella-Garcia M, Shapiro GI, Costa DB, Doebele RC, Le LP, Zheng Z, Tan W, Stephenson P, Shreeve SM, Tye LM, Christensen JG, Wilner KD, Clark JW, Iafrate AJ. Crizotinib in ROS1-rearranged non-small-cell lung cancer. N Engl J Med. 2014 Nov 20;371(21):1963-71. doi: 10.1056/NEJMoa1406766. Epub 2014 Sep 27. PMID 25264305
- [Background] Lennerz JK, Kwak EL, Ackerman A, Michael M, Fox SB, Bergethon K, Lauwers GY, Christensen JG, Wilner KD, Haber DA, Salgia R, Bang YJ, Clark JW, Solomon BJ, Iafrate AJ. MET amplification identifies a small and aggressive subgroup of esophagogastric adenocarcinoma with evidence of responsiveness to crizotinib. J Clin Oncol. 2011 Dec 20;29(36):4803-10. doi: 10.1200/JCO.2011.35.4928. Epub 2011 Oct 31. PMID 22042947
- [Background] Lauren Christine Harshman, K.P.G., Laura Polacek, Mary-Ellen Taplin, Atish Dipankar Choudhury, Mark M Pomerantz, Joaquim Bellmunt, Channing Yu, Zijie Sun, Sandy Srinivas, Philip W. Kantoff, Christopher Sweeney. An investigator-initiated phase I study of crizotinib in combination with enzalutamide in metastatic castration-resistant prostate cancer (mCRPC) before or after progression on docetaxel. in ASCO Annual Meeting. 2016. Chicago: J Clin Oncol.
- [Background] E. L. Kwak, D.R.C., J. Clark, G. I. Shapiro, R. G. Maki, M. J. Ratain, B. Solomon, Y. Bang, S. Ou, R. Salgia. Clinical activity observed in a phase I dose escalation trial of an oral c-met and ALK inhibitor, PF-02341066. in ASCO Annual Meeting. 2009. J Clin Oncol.
- [Background] Di Leo A, Jerusalem G, Petruzelka L, Torres R, Bondarenko IN, Khasanov R, Verhoeven D, Pedrini JL, Smirnova I, Lichinitser MR, Pendergrass K, Garnett S, Lindemann JP, Sapunar F, Martin M. Results of the CONFIRM phase III trial comparing fulvestrant 250 mg with fulvestrant 500 mg in postmenopausal women with estrogen receptor-positive advanced breast cancer. J Clin Oncol. 2010 Oct 20;28(30):4594-600. doi: 10.1200/JCO.2010.28.8415. Epub 2010 Sep 20. PMID 20855825
- [Background] Telford BJ, Chen A, Beetham H, Frick J, Brew TP, Gould CM, Single A, Godwin T, Simpson KJ, Guilford P. Synthetic Lethal Screens Identify Vulnerabilities in GPCR Signaling and Cytoskeletal Organization in E-Cadherin-Deficient Cells. Mol Cancer Ther. 2015 May;14(5):1213-23. doi: 10.1158/1535-7163.MCT-14-1092. Epub 2015 Mar 16. PMID 25777964
- [Background] Al-Batran SE, Homann N, Pauligk C, Goetze TO, Meiler J, Kasper S, Kopp HG, Mayer F, Haag GM, Luley K, Lindig U, Schmiegel W, Pohl M, Stoehlmacher J, Folprecht G, Probst S, Prasnikar N, Fischbach W, Mahlberg R, Trojan J, Koenigsmann M, Martens UM, Thuss-Patience P, Egger M, Block A, Heinemann V, Illerhaus G, Moehler M, Schenk M, Kullmann F, Behringer DM, Heike M, Pink D, Teschendorf C, Lohr C, Bernhard H, Schuch G, Rethwisch V, von Weikersthal LF, Hartmann JT, Kneba M, Daum S, Schulmann K, Weniger J, Belle S, Gaiser T, Oduncu FS, Guntner M, Hozaeel W, Reichart A, Jager E, Kraus T, Monig S, Bechstein WO, Schuler M, Schmalenberg H, Hofheinz RD; FLOT4-AIO Investigators. Perioperative chemotherapy with fluorouracil plus leucovorin, oxaliplatin, and docetaxel versus fluorouracil or capecitabine plus cisplatin and epirubicin for locally advanced, resectable gastric or gastro-oesophageal junction adenocarcinoma (FLOT4): a randomised, phase 2/3 trial. Lancet. 2019 May 11;393(10184):1948-1957. doi: 10.1016/S0140-6736(18)32557-1. Epub 2019 Apr 11. PMID 30982686
- [Background] Bajrami I, Marlow R, van de Ven M, Brough R, Pemberton HN, Frankum J, Song F, Rafiq R, Konde A, Krastev DB, Menon M, Campbell J, Gulati A, Kumar R, Pettitt SJ, Gurden MD, Cardenosa ML, Chong I, Gazinska P, Wallberg F, Sawyer EJ, Martin LA, Dowsett M, Linardopoulos S, Natrajan R, Ryan CJ, Derksen PWB, Jonkers J, Tutt ANJ, Ashworth A, Lord CJ. E-Cadherin/ROS1 Inhibitor Synthetic Lethality in Breast Cancer. Cancer Discov. 2018 Apr;8(4):498-515. doi: 10.1158/2159-8290.CD-17-0603. PMID 29610289
- [Background] Di Leo A, Jerusalem G, Petruzelka L, Torres R, Bondarenko IN, Khasanov R, Verhoeven D, Pedrini JL, Smirnova I, Lichinitser MR, Pendergrass K, Malorni L, Garnett S, Rukazenkov Y, Martin M. Final overall survival: fulvestrant 500 mg vs 250 mg in the randomized CONFIRM trial. J Natl Cancer Inst. 2014 Jan;106(1):djt337. doi: 10.1093/jnci/djt337. Epub 2013 Dec 7. PMID 24317176
- [Derived] Okines A, Irfan T, Asare B, Mohammed K, Osin P, Nerurkar A, Smith IE, Parton M, Ring A, Johnston S, Turner NC. Clinical outcomes in patients with triple negative or HER2 positive lobular breast cancer: a single institution experience. Breast Cancer Res Treat. 2022 Apr;192(3):563-571. doi: 10.1007/s10549-021-06432-z. Epub 2022 Feb 4. PMID 35119530

RESULTS

PARTICIPANT FLOW:
Groups:
- Crizotinib Oral Capsule [Xalkori] Monotherapy: Arm 1 basket (diffuse gastric cancer, triple negative lobular breast cancer and Other CDH1 mutated cancer) cohort
- Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection: Arm 2 ER positive lobular breast cancer cohort
Period: Overall Study
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
Started | 6 | 27
Completed | 6 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Crizotinib Oral Capsule [Xalkori] Monotherapy: Arm 1 - Basket (diffuse gastric cancer, triple negative lobular breast cancer and Other CDH1 mutated cancer) cohort."
- Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection: Arm 2 - ER positive lobular breast cancer cohort
- Total: Total of all reporting groups
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection | Total
Number analyzed (Participants) | 6 | 27 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 21 | 24
  >=65 years | 3 | 6 | 9
Age, Continuous [Median (Full Range); unit: years] | 63 [37 to 83] | 57 [35 to 73] | 57 [35 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 27 | 33
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 27 | 33
Menopausal Status [Count of Participants; unit: Participants]
  Peri-menopausal | 1 | 4 | 5
  Post-menopausal | 4 | 20 | 24
  Pre-menopausal | 1 | 3 | 4
Cancer [Count of Participants; unit: Participants]
  ER positive/HER2 negative Lobular breast cancer | 0 | 27 | 27
  Diffuse gastric cancer | 1 | 0 | 1
  Triple negative lobular breast cancer | 5 | 0 | 5
  other CDH1 Mutated cancer | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Breast Cancer Cohort Participants With Confirmed Response Assessed Using RECIST v1.1
Description: To assess confirmed response rate by RECIST 1.1 of crizotinib and fulvestrant in advanced E-cadherin negative, ER positive lobular breast cancer.
Time Frame: From Day 1 to Progressive Disease, assessed up to end of study (Approximately 57 months)
Population: Patients who receive at least one cycle of the trial medication and had at least one response (RECIST 1.1 scan) post treatment start. Patients who stopped study treatment before the first response evaluation scan has been performed with clinical progression were included in the disease progression category.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
Number analyzed (Participants) | 27
Participants | 1

2. Primary Outcome: Percentage of Basket Cohort Participants With Confirmed Response Assessed Using RECIST v1.1
Description: To assess confirmed response rate (CR/PR outcome) by RECIST 1.1 scan of crizotinib monotherapy in advanced E-cadherin negative, diffuse gastric cancer, triple negative lobular breast cancer or CDH1-mutated solid tumour.
Time Frame: From Day 1 to Progressive Disease, assessed up to end of study (Approximately 57 months)
Population: Patients who received at least one cycle of the trial medication and had at least one response (RECIST 1.1 scan) post treatment start. Patients who stopped study treatment before the first response evaluation scan has been performed with clinical progression were included in the disease progression category.
Measure: Count of Participants; unit: Participants
Groups:
- Crizotinib Oral Capsule [Xalkori] Monotherapy: Arm 1 - Basket (diffuse gastric cancer, triple negative lobular breast cancer and Other CDH1 mutated cancer) cohort.
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: To assess the overall safety and tolerability of crizotinib with fulvestrant in the breast cancer cohort and as monotherapy in the basket cancer cohort. Toxicity will be assessed by CTCAE (version 4) every 4 weeks during study treatment. Adverse events, including serious adverse events, will be recorded until 30 days after the last dose of study treatment with crizotinib.
Time Frame: From Day 1 to 30 days after last dose of study drug, assessed up to end of study (Approximately 57 months)
Population: Intention to treat (ITT) analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
Number analyzed (Participants) | 6 | 27
Participants | 6 | 27

4. Secondary Outcome: Progression-free Survival (PFS) Assessed Using Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in Both Basket and Breast Cancer Cohorts
Description: PFS is defined as the time from baseline treatment to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first. PD is defined as greater than or equal to (>/=) 20 percent (%) relative increase and >/=5 millimeter (mm) of absolute increase in the sum of diameters (SD) of target lesions (TLs), taking as reference the smallest SD recorded since treatment started, or appearance of 1 or more new lesions.
Time Frame: From Day 1 to disease progression (PD) or death from any cause, assessed up to end of study (Approximately 57 months)
Population: Intention to treat (ITT) analysis population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
Number analyzed (Participants) | 6 | 27
months | 1.8 [0.5 to NA] — The upper boundary of the 95% confidence interval of the PFS not estimable due to small number of subjects recruitment and events observed. | 1.8 [1.1 to 3.2]

5. Secondary Outcome: Assessment of Overall Survival in Each Cohort
Description: Overall survival, calculated from day 1 of study treatment to the date of death from any cause.
Time Frame: From Day 1 to disease progression (PD) or death from any cause, assessed up to end of study (Approximately 57 months)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
Number analyzed (Participants) | 6 | 27
months | 4.4 [1.3 to NA] — The upper boundary of the 95% confidence interval of the OS not estimable due to the small number of subjects recruitment and events observed. | 17.5 [6.9 to 26.0]

ADVERSE EVENTS:
Time Frame: For eligible patients, serious adverse event (SAE) and adverse event (AE) collection commenced from Day 1 (at the time the first patient provided their written informed consent to participate in the trial) and continued until 30 days after the last administration of study drug, assessed up to end of study (approximately 57 months)
Groups:
- Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection: Arm 2 - ER positive lobular breast cancer
Arm/Group | Crizotinib Oral Capsule [Xalkori] Monotherapy | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection
All-Cause Mortality (participants affected / at risk) | 6/6 | 20/27
Serious Adverse Events (participants affected / at risk) | 4/6 | 5/27
Other Adverse Events (participants affected / at risk) | 6/6 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib Oral Capsule [Xalkori] Monotherapy (N=6) | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection (N=27)
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 1
Fever (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Crizotinib Oral Capsule [Xalkori] Monotherapy (N=6) | Crizotinib Oral Capsule [Xalkori] Plus Fulvestrant Injection (N=27)
Alanine aminotransferase increased (Investigations) | 4 | 17
Aspartate aminotransferase increased (Investigations) | 4 | 20
Abdominal pain (Gastrointestinal disorders) | 2 | 8
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 10
Gastrointestinal pain (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 16
Edema trunk (General disorders) | 2 | 0
Creatinine increased (Investigations) | 2 | 4
Lymphocyte count decreased (Investigations) | 2 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 4
Dysgeusia (Nervous system disorders) | 2 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 12
Flashing lights (Eye disorders) | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 1 | 3
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 13
Nausea (Gastrointestinal disorders) | 1 | 20
Obstruction gastric (Gastrointestinal disorders) | 1 | 0
Edema limbs (General disorders) | 1 | 3
Fatigue (General disorders) | 1 | 12
Pain (General disorders) | 1 | 2
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0
Alkaline phosphatase increased (Investigations) | 1 | 9
Anorexia (Metabolism and nutrition disorders) | 1 | 3
Hyponatremia (Metabolism and nutrition disorders) | 1 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Other (Blood and lymphatic system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 0 | 8
GGT increased (Investigations) | 0 | 6
Headache (Nervous system disorders) | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Blurred vision (Eye disorders) | 0 | 5
Neutrophil count decreased (Investigations) | 0 | 5
Sinus bradycardia (Cardiac disorders) | 0 | 4
Fever (General disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 0 | 3
Flu like symptoms (General disorders) | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 2
Platelet count decreased (Investigations) | 0 | 3
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 2
Bloating (Gastrointestinal disorders) | 0 | 2
Localized edema (General disorders) | 0 | 2
White blood cell decreased (Investigations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Paresthesia (Nervous system disorders) | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hot flashes (Vascular disorders) | 0 | 2
Hypertension (Vascular disorders) | 0 | 2
Other (Eye disorders) | 0 | 4
Other (Gastrointestinal disorders) | 2 | 3
Other (General disorders) | 3 | 7
Other (Infections and infestations) | 0 | 2
Other (Investigations) | 0 | 6
Other (Musculoskeletal and connective tissue disorders) | 1 | 2
Other (Nervous system disorders) | 0 | 2
Other (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Other (Skin and subcutaneous tissue disorders) | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/43/NCT03620643/Prot_SAP_000.pdf